CLINICAL TRIAL: NCT04551560
Title: Stress and Congestive Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2000027107; 1R01HL152548-01 (NIH)
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mental Stress (Other): Patients will undergo a lab mental stress protocol, and a field protocol using ecological momentary assessment (EMA) to test the effects of psychological stress and negative emotion on PAP in HF patients.
  Interventions: Other: Mental Stress

INTERVENTIONS:
Other: Mental Stress — Patients will undergo a lab mental stress protocol, and a field protocol using ecological momentary assessment (EMA) to test the effects of psychological stress and negative emotion on PAP in HF patients.

SUMMARY:
The purpose of this study is to investigate whether acute stress can precipitate congestive heart failure (CHF) exacerbation in patients with CHF.

DETAILED DESCRIPTION:
Study participants will be followed for 6 months. Patients will undergo a laboratory mental stress protocol, and a field protocol using ecological momentary assessment (EMA) to, 1) test the effects of psychological stress and negative emotion on pulmonary artery pressure (PAP) in HF patients; 2) examine the relationship of stress-induced PAP change to HF exacerbation; and 3) identify a risk profile by exploring predictors of heterogeneity in the PAP response to stress, including physiological variables (e.g., NYHA class, biomarkers), sleep, quality, and psychosocial variables (e.g., sources of chronic stress, anger/hostility, depression. Patients will also undergo a battery of psychosocial questionnaires either online or paper as they prefer.

Laboratory Component HF patients with existing or newly implanted with a CardioMEMS PAP monitor will complete the laboratory stress protocol, in the Hospital Research Unit (HRU) or other YCCI outpatient sites. Resting quiet period (30 min) Relaxation (10min) Stress period (10min) Recovery (30min) follows the stress task followed by Neutral conversation (5min). PAP and blood pressure are assessed, and the participant completes a stress/mood likert assessment at the end of the rest period, stress, and 15min and 30min during recovery.

Blood drawing: 10 ml of blood will be drawn for a panel of CHF-related biomarkers either at the beginning of the laboratory session or in a clinic visit and 1 vial drawn at the end of rest, stress and twice during recovery.

Field Component: For this phase, they will complete PAP assessment in the morning for six months, following their standard clinical protocol for daily monitoring (standard of care). In addition, at the time of the morning PAP assessment they will complete eDiary-based EMA via likert style questions (e.g., on an anchored, 1-100 scale) concerning the quality of their sleep the night before, the level of stress they are currently experiencing, and their emotional state. For one month, they will complete an additional evening PAP assessment, (extra, not standard of care) at which time they will complete similar eDiary-based likert style questions concerning the stressfulness of their day and the sources of stress (if any) they have experienced. All questions will be completed using the smartphone based EMA 'app' that the team has used and are currently using in NIH funded studies.

Follow up - Clinical outcomes will be determined through review of the Cardiomems Merlin database and medical record review & Baseline psychosocial questionnaires.

ELIGIBILITY:
Inclusion Criteria:

-Heart failure patients over 18 who have or will be receiving a Cardiomems implanted PAP monitor.

Exclusion Criteria:

* Patients who are unable to perform EMA or laboratory assessments due to cognitive, visual, language, or other disabilities will be excluded.
* Patients with Class IV heart failure will also be excluded, as they are already maximally decompensated, and a ceiling/floor effect would preclude effects of stress.
* Patients with conditions other than heart failure that affect PA pressures (e.g. dialysis).
* Patients with physical conditions that interfere with study participation.
* Patients non-compliant with their PAP monitoring.
* Patients with chronic opioid use will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2020-12-02 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Artery Pressure | 6 months
  Pulmonary artery pressure as measured by an implanted monitor: Pulmonary artery pressure will be compared between times of stress and calm, in both the laboratory and real-life setting.

SECONDARY OUTCOMES:
Medication changes | 6 months
  Will be compared between those with highest levels of stress-triggered PA increases, and those with lower

OTHER OUTCOMES:
Number of participants that are hospitalized | 6 months
  Hospitalizations will be compared between those with highest levels of stress-triggered PA increases, and those with lower

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Lampert, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - St. Francis Hospital, Hartford, Connecticut
  - Yale University, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No